CLINICAL TRIAL: NCT06221722
Title: Evaluation of Brain Connectivity Function in Predicting Therapeutic Effects in Patients With Refractory Constipation: a Multicenter, Prospective, Cohort Study
Brief Title: Predicting Treatment Outcomes in Refractory Constipation Through Brain Connectivity Evaluation
Status: Recruiting | Type: Observational
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Zhifeng Zhao, PhD, Dr., Xijing Hospital of Digestive Diseases
Other Study IDs: KY20232332-C-1
Record Dates: First submitted 2023-12-26; First posted 2024-01-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Constipation - Functional; Refractory Constipation; Fluoxetine; fMRI; Brain Connectivity; Treatment Efficacy; Somatic Symptom; Mental Symptom
Keywords: fMRI; functional connectivity; refractory constipation
MeSH Terms: conditions — Constipation; Medically Unexplained Symptoms | interventions — Fluoxetine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool, Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Refractory constipation: fluoxetine sensitive: Functional constipation patients maintained at least 3 months of continuous regular therapy with ineffective treatment. The treatment included the utilization of osmotic laxatives, stimulant laxatives, prosecretory agents, and a high-fibre diet.
  After 3 months of regular treatment, patients received fluoxetine therapy for 4-week with effective treatment of constipation symptoms.
  Interventions: Diagnostic Test: BOLD-fMRI; Drug: Regular treatment of functional constipation; Drug: fluoxetine
- Refractory constipation: fluoxetine insensitive: Functional constipation patients maintained at least 3 months of continuous regular therapy with ineffective treatment. The treatment included the utilization of osmotic laxatives, stimulant laxatives, prosecretory agents, and a high-fibre diet.
  After 3 months of regular treatment, patients received fluoxetine therapy for 4-week with ineffective treatment of constipation symptoms.
  Interventions: Diagnostic Test: BOLD-fMRI; Drug: Regular treatment of functional constipation; Drug: fluoxetine
- Non-refractory constipation: Functional constipation patients maintained at least 3 months of continuous regular therapy with effective treatment. The treatment included the utilization of osmotic laxatives, stimulant laxatives, prosecretory agents, and a high-fibre diet.
  Interventions: Diagnostic Test: BOLD-fMRI; Drug: Regular treatment of functional constipation
- Health Control: Volunteers without symptoms of constipation
  Interventions: Diagnostic Test: BOLD-fMRI

INTERVENTIONS:
Diagnostic Test: BOLD-fMRI — Blood-Oxygen-Level Dependent Functional Magnetic Resonance Imaging
Drug: Regular treatment of functional constipation — at least 3 months of continuous regular treatment. This treatment included the utilization of osmotic laxatives, stimulant laxatives, prosecretory agents, and a high-fibre diet.
  Groups: Non-refractory constipation; Refractory constipation: fluoxetine insensitive; Refractory constipation: fluoxetine sensitive
Drug: fluoxetine — Fluoxetine oral treatment for 4 weeks.
  Groups: Refractory constipation: fluoxetine insensitive; Refractory constipation: fluoxetine sensitive

SUMMARY:
The goal of this observational study is to identify the characteristics of brain functional connectivity in refractory constipation and fluoxetine-sensitive patients. The main questions it aims to answer are:

* Investigating the alterations in brain functional connectivity in patients with refractory constipation and fluoxetine-sensitive patients
* Assessing the predictive value of brain functional connectivity regarding the efficacy of fluoxetine and standard protocol treatments for constipation.

Participants will receive:

* Standard physiological and psychological assessments of constipation
* BOLD-fMRI tests
* Standard protocol and fluoxetine treatment

If there is a comparison group: Researchers will compare:

Refractory group/Fluoxetine sensitive group to see the specific brain alterations.

ELIGIBILITY:
Inclusion Criteria:

* 18≤ age ≤ 45 years old
* Right-handed
* Patients diagnosed as functional constipation according to the Rome IV criteria
* Informed consent of patients

Exclusion Criteria:

* Complicated with gastrointestinal organic disease or significant functional abnormalities (tuberculosis, polyps, Crohn's disease, tumors, congenital megacolon, pelvic floor muscle relaxation, abnormal colonic transit test, etc.)
* Long-term intense exercise (continuous exercise for more than 8 hours per week, such as marathon runners or triathletes)
* No history of chronic pain, no recent major trauma
* Drug abuse or tobacco dependence (half a pack or more per day)
* Combined hypothyroidism and Parkinson's disease
* Patients with confirmed mental illness or neurological disorders who take psychotropic drugs, analgesics or hormones
* History of abdominal surgery (appendectomy, hysterectomy, or cholecystectomy)
* Contraindications to functional magnetic resonance imaging (claustrophobia, metal implants)
* Pregnant or lactating women with constipation after delivery
* Patients with other benign and malignant tumors and autoimmune diseases
* Infectious diseases such as hepatitis B, hepatitis C, AIDS, etc.
* Heart disease, organ failure and other chronic diseases that require long-term medication or affect the quality of life

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: tertiary hospitals received patients from northwest of China
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Brain functional connectivity changes in BOLD-fMRI examination in refractory constipation before and after fluoxetine treatment | 1-week pre and 4-week post of fluoxetine treatment
  BOLD-fMRI tests before and after fluoxetine treatment

SECONDARY OUTCOMES:
Changes in PAC-QOL self-assessment scores from baseline | 1-week pre and 4-week post-fluoxetine treatment.
  The Patient Assessment of Constipation Quality of Life (PAC-QOL) questionnaire is a self-reported instrument designed to measure the quality of life in individuals with constipation. This tool comprises 28 items across four fundamental domains, including physical discomfort, worries and concerns, psychosocial discomfort, and satisfaction. In our study, the Chinese version (version 16) was utilized.
Changes in PHQ-15 self-assessment scores relative to baseline. | 1-week pre and 4-week post-fluoxetine treatment.
  The Patient Health Questionnaire-15 (PHQ-15) is a self-reporting inventory that evaluates the severity of somatic symptoms in patients. Comprising 15 items, the questionnaire primarily focuses on experienced bodily symptoms and aids healthcare providers in identifying potential somatization disorders or severe somatic illnesses.
Changes in GAD-7 self-assessment scores from baseline. | 1-week pre and 4-week post-fluoxetine treatment.
  The Generalized Anxiety Disorder-7 (GAD-7) is a brief measure assessing the frequency of anxiety symptoms over the past two weeks. With 7 items, the scale concentrates on the core symptoms of generalized anxiety disorder, serving as an instrument to ascertain the level of anxiety and to monitor the improvement of anxiety symptoms.
Changes in PHQ-9 self-assessment scores since baseline. | 1-week pre and 4-week post-fluoxetine treatment.
  The Patient Health Questionnaire-9 (PHQ-9) is a tool used for screening, diagnosing, monitoring, and quantifying the severity of depression. The questionnaire consists of 9 items drawing from typical symptoms of depression, facilitating the evaluation of the presence and severity of depression by medical professionals.
Changes in KESS self-assessment scores from baseline. | 1-week pre and 4-week post-fluoxetine treatment.
  The KESS questionnaire, Kovacs' Evaluation of Sphincter Symptoms, is utilized to assess defecatory dysfunction. It includes a series of items that inquire about constipation symptoms and defecatory habits, aiming to evaluate the severity and impact of a patient's defecatory disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Qingchuan Zhao, Prof., Study Chair — Xijing Hospital of Digestive Diseases
Locations (3):
- China (3):
  - People's Hospital of Ningxia Hui Autonomous Region, Yinchuan, Ningxia
  - Xi'an International Medical Center Hospital, Xi'an, Shaanxi
  - Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: Yes
Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact zhaozhifeng@outlook.com.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: For more information or to submit a request, please contact zhaozhifeng@outlook.com.
URL: https://prsinfo.clinicaltrials.gov/definitions.html